CLINICAL TRIAL: NCT00691275
Title: Ondansetron vs. Placebo in the Management of Children With Dehydration Due to Acute Gastroenteritis
Brief Title: Efficacy Study of IV Fluids Only vs Ondansetron to Treat Dehydration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sam Reid, MD, Children's Hospitals and Clinics of Minnesota
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0801-012
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Dehydration; Gastroenteritis
Keywords: dehydration; acute gastroenteritis; ondansetron; rehydration
MeSH Terms: conditions — Dehydration; Gastroenteritis | interventions — Ondansetron; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Saline
  Interventions: Drug: Saline
- 1 (Active Comparator): Zofran
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron
  Arms: 1
Drug: Saline
  Arms: 2

SUMMARY:
Dehydration due to vomiting is a common complication of acute gastroenteritis in children. Persistent vomiting following rehydration is a problem in outpatient management using oral rehydration therapy.

Four previous studies have examined the role of the medication, ondansetron, in treating nausea and vomiting in children with gastroenteritis and have suggested that it may be beneficial [1-4]. A previous study has also shown that the administration of intravenous fluid alone to children with dehydration due to gastroenteritis helps resolve nausea and vomiting in the majority of patients [5]. None of the previous studies compared the efficacy of intravenous ondansetron with that of intravenous fluid alone in the prevention of vomiting . In addition, the previous studies were limited by poorly defined inclusion criteria and outcome measures.

The proposed study seeks to more clearly define the role of intravenous ondansetron in the management of children suffering dehydration due to acute gastroenteritis. If ondansetron further reduces the incidence of vomiting compared with intravenous fluid alone, more children with dehydration due to acute gastroenteritis may be successfully discharged to home from the emergency department instead of admitted to the hospital. If it does not, the widespread use of ondansetron for such patients could be discouraged and money could be saved.

Hypothesis:

Patients receiving ondansetron in addition to intravenous fluids for the treatment of dehydration due to vomiting caused by gastroenteritis will not have a significant reduction in the occurrence of persistent vomiting as compared to those who receive only intravenous fluids.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months - 5 years
* Clinical diagnosis of acute gastroenteritis
* Mild or moderate dehydration as determined by validated clinical scale
* Clinical assessment to begin IV fluids
* Vomiting ≥ 2 episodes in past 4 hours

Exclusion Criteria:

* Severe dehydration
* History of significant gastrointestinal, metabolic, renal or cardiac disorder
* Ondansetron allergy
* Non-English language proficient parent/guardian
* Parent/guardian has no telephone

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Received further IV fluids | 2-7 days post discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sam Reid, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota; Henry Ortega, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota; Jeffrey Louie, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota

REFERENCES:
- [Background] Freedman SB, Adler M, Seshadri R, Powell EC. Oral ondansetron for gastroenteritis in a pediatric emergency department. N Engl J Med. 2006 Apr 20;354(16):1698-705. doi: 10.1056/NEJMoa055119. PMID 16625009
- [Background] Reeves JJ, Shannon MW, Fleisher GR. Ondansetron decreases vomiting associated with acute gastroenteritis: a randomized, controlled trial. Pediatrics. 2002 Apr;109(4):e62. doi: 10.1542/peds.109.4.e62. PMID 11927735
- [Background] Ramsook C, Sahagun-Carreon I, Kozinetz CA, Moro-Sutherland D. A randomized clinical trial comparing oral ondansetron with placebo in children with vomiting from acute gastroenteritis. Ann Emerg Med. 2002 Apr;39(4):397-403. doi: 10.1067/mem.2002.122706. PMID 11919526
- [Background] Stork CM, Brown KM, Reilly TH, Secreti L, Brown LH. Emergency department treatment of viral gastritis using intravenous ondansetron or dexamethasone in children. Acad Emerg Med. 2006 Oct;13(10):1027-33. doi: 10.1197/j.aem.2006.05.018. Epub 2006 Aug 10. PMID 16902049
- [Background] Reid SR, Bonadio WA. Outpatient rapid intravenous rehydration to correct dehydration and resolve vomiting in children with acute gastroenteritis. Ann Emerg Med. 1996 Sep;28(3):318-23. doi: 10.1016/s0196-0644(96)70032-x. PMID 8780476